CLINICAL TRIAL: NCT00676273
Title: TVT-Secur Versus TVT-Obturator: A Randomized Trial of Suburethral Sling Operative Procedures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Urogynecology Associates (Other)
Responsible Party: Peter Rosenblatt, MD, Boston Urogynecology Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28142
Record Dates: First submitted 2007-11-16; First posted 2008-05-13 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): TVTO
  Interventions: Device: TVT-Obturator (TVT-O)
- 2 (Active Comparator): TVTS
  Interventions: Device: TVT-Secur (TVT-S) (Hammock method)

INTERVENTIONS:
Device: TVT-Obturator (TVT-O) — sub urethral sling
  Arms: 1
Device: TVT-Secur (TVT-S) (Hammock method) — suburethral sling
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether TVT-Secur (TVT-S) (Hammock method) and TVT-Obturator (TVT-O) suburethral sling procedures have equivalent patient satisfaction and clinical efficacy in the treatment of stress urinary incontinence alone or the stress component in mixed urinary incontinence.

DETAILED DESCRIPTION:
Patient satisfaction will be measured by symptom quality of life questionnaires (pre-operatively, 3 months and one year) and patient pain will be measured by verbal analogue rating scale (post-operative day 1 and day 7). Clinical efficacy will be measured by a cough stress test pre-operatively and post-operatively at 3 months and 1 year. A Q-tip test will also be performed pre-operatively and at 3 months and 1 year post-operatively. Subjects will be followed for a minimum of one year to evaluate recurrence of symptoms and complications, including the rate of mesh erosion, time to normal void in the post-operative period, the rate of sling revision, post-operative pain, voiding dysfunction and de novo urgency.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age
* Demonstrate a positive cough stress test during complex multi-channel urodynamic testing
* Demonstrate impact of stress urinary incontinence on quality of life questionnaire
* Are able to comprehend and sign a written informed consent
* Understand and are willing to comply with the study requirements, including agreeing to be available for the follow-up evaluations
* Are psychologically stable and suitable for interventions determined by the investigator
* Are ambulatory and able to use a toilet independently

Exclusion Criteria:

Patients:

* Who are pregnant or planning to become pregnant during the study or in the future
* With a elevated post-void residual (defined as PVR > 100cc)
* With a bleeding condition or on anti-coagulant therapy
* With immunosuppression (i.e. HIV, lymphoma)
* With multiple sclerosis or other progressive neurological disease
* With evidence of a local or systemic infection, including urinary tract infection
* With evidence of intrinsic sphincter deficiency as defined by a maximal urethral closure pressure of <20 cm H2O
* Previous sub-urethral sling
* Predominant overactive bladder symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-03 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of TVT-S versus TVT-O suburethral slings in the treatment of stress urinary incontinence or the stress incontinence component of mixed urinary incontinence by the presence or absence or urinary incontinence on cough stress test. | 1 year

SECONDARY OUTCOMES:
To describe or assess known side effects or complications,post-operative pain, time of return to daily activities of living, improvement in patient quality of life, change in Q-tip test | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rosenblatt, MD, Principal Investigator — Boston Urogynecology Associates; Lekha Hota, MD, Study Director — Boston Urogynecology Associates
Locations (1):
- Boston Urogynecology Associates, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839